CLINICAL TRIAL: NCT02014623
Title: Immunological Mechanisms of Oralair® (5 Grass Mix Sublingual Allergen Immunotherapy Tablet) in Patients With Seasonal Allergic Rhinitis
Brief Title: Immunological Mechanisms of Oralair® in Patients With Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 514/13
Record Dates: First submitted 2013-11-19; First posted 2013-12-18 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis; Asthma; Regulatory T cells; IgE; IgG4
MeSH Terms: conditions — Rhinitis, Allergic; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grass pollen sublingual immunotherapy tablet (Active Comparator): A sublingual allergen immunotherapy tablet (Oralair) containing: 300 index of reactivity (IR) of 5 grass pollen allergen extracts:perennial ryegrass (Lolium perenne), meadow grass (Poa pratensis), timothy grass (Phleum pratense), cocksfoot (Dactylis glomerata) and sweet vernal grass (Anthoxanthum odoratum) in an open label fashion administered for 4 months prior to the pollen season.
  Interventions: Other: Grass pollen sublingual immunotherapy tablet
- Control (Other): Standard medical therapy: oral antihistamines AND/OR nasal steroids AND/OR nasal antihistamines
  Interventions: Drug: Control

INTERVENTIONS:
Other: Grass pollen sublingual immunotherapy tablet
  Arms: Grass pollen sublingual immunotherapy tablet
Drug: Control
  Other Names: Oral anthistamines AND/OR Nasal steroids AND/OR Nasal antihistamines
  Arms: Control

SUMMARY:
Allergic diseases represent a major health issue worldwide and epidemiological studies in Melbourne, Australia, have reported a high prevalence of rhinitis (hayfever) and atopy (genetic tendency to make allergy antibody) in Asian and Caucasian subjects. Mainstay treatment of allergic rhinitis is allergen avoidance and pharmacotherapy for symptom relief. Allergen immunotherapy offers the advantages of specific treatment with long lasting efficacy, and can modify the course of disease. However, use of this treatment is restricted by the high risk of adverse events especially in asthmatics. Other, better tolerated, routes of allergen administration than the current conventional subcutaneous route (SCIT) have been investigated including the sublingual route (SLIT) and recently sublingual tablets for pollen allergy immunotherapy became available. The tablets are safe and easy to use and contain pollen extracts from 5 of the most common allergy-causing European grasses but include ryegrass (Lolium perenne), the major seasonal pollen for allergy in Melbourne and south-eastern Australia. The immunological mechanisms of sublingual immunotherapy are not fully understood. The investigators propose conducting a longitudinal open label study to investigate the immunological changes that occur with the 5 grass pollen sublingual immunotherapy tablet (Oralair®) in a cohort of Chinese and non-Chinese background subjects. The investigators will investigate the induction of relevant T cell regulatory immune mechanisms and changes in serum allergen-specific immunoglobulin (Ig) E and IgG4. Immunoregulatory cytokine synthesis and T cell phenotype (Bio-plex and flow cytometry) will be examined. This project will provide important fundamental knowledge on which to inform decisions for the greater application of this treatment for subjects with moderate and severe allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of Chinese heritage or non-Chinese heritage
* Clinical diagnosis of moderate to severe seasonal allergic rhinitis
* Ryegrass-specific IgE : CAP-Pharmacia score > 1

Exclusion Criteria:

* Ongoing immunotherapy or previous immunotherapy (within last 5 years)
* Continuous oral corticosteroids
* Moderate, severe or unstable asthma
* Standard contraindications for allergen immunotherapy
* Ongoing treatment with β-blockers
* Immunodeficiency diseases
* Malignancy
* Significant inflammatory condition or disease in the oral cavity

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Ryegrass specific-IgG4 at 4 months and 12 months | Baseline, 4 months, 12 months

SECONDARY OUTCOMES:
Change in Quality of Life assessed by an Allergic Rhinitis Quality of Life Questionnaire at 4, 8 and 12 months | Baseline, 4 months, 8 months, 12 months
Change in Combined Symptoms and Medication requirements score at 4, 8 and 12 months | Baseline, 4 months, 8 months, 12 months
Change in Fractional Exhaled Nitric Oxide at 4, 8, and 12 months | Baseline, 4 months, 8 months, 12 months
Change in Helper and regulatory T cell response to ryegrass pollen at 4 months and 12 months | Baseline,4 months, 12 months
Change in Ryegrass-specific IgE at 4 months and 12 months | Baseline, 4 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robyn O'Hehir, MBBS MBBS FRACP FRCP PhD, Principal Investigator — Director, Department of Allergy, Immunology and Respiratory Medicine, The Alfred Hospital; Mark Hew, MBBS FRACP PhD, Study Director — Head of Allergy, Asthma and Clinical Immunology Service, Department of Allergy, Immunology and Respiratory Medicine, The Alfred Hospital; Jennifer Rolland, BSc, PhD, Study Chair — Emeritus Professor Central Clinical School Monash University; Alessandra Sandrini, MD, PhD, Study Chair — Senior Clinical Fellow, Department of Allergy, Immunology and Respiratory Medicine, The Alfred Hospital; Celia Zubrinich, MBBS FRACP, Study Chair — Consultant, Department of Allergy, Immunology and Respiratory Medicine, The Alfred Hospital; Nirupama Varese, BSc Hons, MSc, Study Chair — Research Officer, Central Clinical School Monash University
Locations (1):
- Department of Allergy, Immunology and Respiratory Medicine, The Alfred Hospital- Bayside Health, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] O'Hehir RE, Varese NP, Deckert K, Zubrinich CM, van Zelm MC, Rolland JM, Hew M. Epidemic Thunderstorm Asthma Protection with Five-Grass Pollen Tablet Sublingual Immunotherapy: A Clinical Trial. Am J Respir Crit Care Med. 2018 Jul 1;198(1):126-128. doi: 10.1164/rccm.201711-2337LE. No abstract available. PMID 29461859